CLINICAL TRIAL: NCT05448482
Title: Hybrid Versus Synthetic Transobturator Tape for Treatment of Female Stress Urinary Incontinence: Prospective Randomised Study
Brief Title: Hybrid Versus Synthetic TOT for Treatment of SUI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Serial No : 0202538
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-03

CONDITIONS: Female Stress Incontinence
MeSH Terms: interventions — Suburethral Slings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid transobturator tape (Experimental): Anterior rectus fascia will be exposed and an approximately 8-10 cm × 1 cm strip of rectus fascia will be marked out. The sling will be harvested using sharp dissection. Thereafter, a Polyprolene monofilamentous mesh of 15 cm x 1 cm will be sutured to each edge of the rectus fascia sling that had been harvested.
  Then, a 2-cm midline incision over the anterior vaginal wall at the level of mid-urethra. A combination of blunt and sharp dissection will be carried out to the obturator foramen bilaterally.
  Next, a stab incision will be made at a point approximately 2.5 cm infero-lateral to the pubic tubercle bilaterally, corresponding to the level of clitoris. A trocar will be passed through each obturator foramen (outside-in) and the edge of the mesh will be retracted through the incision. Next, the retraction of both meshes will continue until the rectus fascia sling remain flushed with the urethra.
  Interventions: Procedure: Transobturator tape
- Conventional transobturator tape (Active Comparator): The conventional mesh using mid urethral sling through the trans obturator route
  Interventions: Procedure: Transobturator tape

INTERVENTIONS:
Procedure: Transobturator tape — Mid urethral sling for treatment of female stress urinary incontinence

SUMMARY:
This prospective study is conducted on female patients presenting with SUI at Alexandria main university hospital. Patients with neurogenic voiding dysfunction, history of anti-incontinence surgery, urge-predominant MUI, urogenital cancer, pelvic irradiation, body mass index more than 40 kg/m2 and more than stage 1 POP are excluded. Patients are randomized into 2 groups, one group will be subjected to h_TOT, and the second group to conventional TOT. Patients are subjected to PGI and UDI-6 questionnaires and a urodynamic study before and 6 months after the both surgery. Success is defined as: no subjective complaint of SUI, negative cough stress test and no leakage on UDS.

DETAILED DESCRIPTION:
The present study will be a single center randomized clinical trial. Recruitment will be performed among women presented to Alexandria Main University Hospital urology clinic complaining of urinary stress incontinence, in whom surgery was regarded as the treatment of choice.

Women will be eligible if they have a positive stress test. The stress test will be performed in a semi lithotomy position with a semi full bladder. Women will be randomized into the groups by using Sealed Opaque Envelope System. Patients will be randomized into 2 groups of 25 patient each. One group will be subjected to hybrid TOT, and the second to conventional TOT.

Preoperative and post-operative (at 3 and 6 months) will include:

* Clinical examination including cough stress test.
* Patient global impression questionnaire (PGI)
* Patient questionnaire for incontinence (UDI-6)
* Urodynamic (pressure-flow study)

No concomitant surgery will be performed on women enrolled in the trial. All patients will give a written informed consent.

Technique of hybrid TOT The procedure will be performed while the patient is in dorsal lithotomy position under spinal saddle anesthesia.

A sterile 14 Fr. Foley catheter will be placed per urethra to empty the bladder. The next step will be to harvest a strip of rectus fascia. A 4-5 cm transverse abdominal incision will be made 2 cm cephalad to the pubic symphysis. Anterior rectus fascia will be exposed and an approximately 8-10 cm × 1 cm strip of rectus fascia will be marked out. The sling will be harvested using sharp dissection and the anterior rectus fascia defect will be reapproximated using 1-0 Prolene suture. Thereafter, a Polyprolene monofilamentous mesh of 15 cm x 1 cm will be sutured to each edge of the rectus fascia sling that had been harvested.

Then, normal saline will be injected in the space between the anterior vaginal wall and mid urethra for hydrodissection, followed by a 2-cm midline incision over the anterior vaginal wall at the level of mid-urethra. A combination of blunt and sharp dissection will be carried out to the obturator foramen bilaterally.

Next, a stab incision will be made at a point approximately 2.5 cm infero-lateral to the pubic tubercle bilaterally, corresponding to the level of clitoris. A trocar (C-shaped, specially built for the TOT) will be passed through each obturator foramen (outside-in) and the edge of the mesh will be retracted through the incision. The same process will be repeated on the other side. Next, the retraction of both meshes will continue until the rectus fascia sling remain flushed with the urethra. An artery forceps will be kept between the fascia and the urethra to avoid excessive tension. Excess mesh on each side will be removed.

The sling will be secured to the peri-urethral tissue with interrupted polyglactin 4-0 suture to prevent rolling and to ensure a flat, broad based sling. The stab incisions will be closed. The anterior vaginal wall will be closed with polyglactin 4-0 suture. Vagina will be packed with povidone iodine-soaked gauze. Vaginal pack and urethral catheter will be removed in the morning of the first postoperative day.

The 2 groups will be compared using the standard statistical methods regarding outcomes and complications. The primary outcome of the study will be achievement of continence (efficacy) while the secondary outcomes will include intraoperative and early post-operative complications, convalescence, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Clinically proven SUI or stress-predominant mixed urinary incontinence by cough stress test.

Exclusion Criteria:

* • Patients with neurogenic voiding dysfunction.

  * History of anti-incontinence surgery.
  * Presence of urge-predominant mixed urinary incontinence.
  * Peripheral neuropathy.
  * Multiple sclerosis.
  * History of urogenital cancer.
  * Pelvic irradiation
  * Body mass index more than 40 kg/m2
  * The presence of more than stage 2 pelvic organ prolapse as per pelvic organ prolapse quantification (POP-Q) system score.
  * Active urinary tract infection
  * Pregnant women

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2023-01-05 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
Dryness | 6 months
  Absence of clinical and urodynamic stress incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No